CLINICAL TRIAL: NCT05934110
Title: A 26-week, Double-blind, Randomized Study in Participants With Overweight or Obesity Investigating the Added Contribution of Acarbose in EMP16 on Efficacy, Safety and Tolerability
Brief Title: Study Exploring the Supportive Effect of Acarbose in Weight Management
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Empros Pharma AB (Industry)
Collaborators: CTC Clinical Trial Consultants AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EP-003; 2022-003320-40 (EudraCT Number)
Record Dates: First submitted 2023-05-29; First posted 2023-07-06 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Overweight or Obesity
Keywords: Overweight, Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Orlistat

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind study in participants with overweight or obesity in which the effect of acarbose and the impact of dose on efficacy, safety and tolerability is investigated by comparing the EMP16 combination product with modified release (MR) orlistat, orlistat in its conventional dosage form and placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study, and the allocation of treatments will not be disclosed until clean file has been declared and the database has been locked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- EMP16-120/40 (Experimental): EMP16 120 mg orlistat/40 mg acarbose (referred to as EMP16-120/40), 80 participants.
  Interventions: Drug: EMP16-120/40
- MR orlistat (Active Comparator): MR orlistat 120 mg, 80 participants.
  Interventions: Drug: MR orlistat 120 mg
- Conventional orlistat (Active Comparator): Conventional orlistat 120 mg, 80 participants.
  Interventions: Drug: Conventional orlistat 120 mg,; Drug: Placebo
- EMP16-60/20 (Experimental): EMP16 60 mg orlistat/20 mg acarbose (referred to as EMP16-60/20), 40 participants.
  Interventions: Drug: EMP16-60/20; Drug: Placebo
- Placebo (Placebo Comparator): Placebo, 40 participants
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EMP16-120/40 — EMP16 is supplied as oral MR capsules with the strength of 60 mg orlistat/20 mg acarbose.
  Dosage:
  week 1-2: 60 mg orlistat/20 mg acarbose (1 capsule per day), week 3-4: 60 mg orlistat/20 mg acarbose (1 capsule TID), week 5-26: 60 mg orlistat/20 mg acarbose (2 capsules TID).
  Arms: EMP16-120/40
Drug: MR orlistat 120 mg — MR orlistat 120 mg is the same as EMP16-120/40 but without the acarbose component in matching oral capsules.
  Dosage:. week 1-2: 60 mg MR orlistat (1 capsule per day), week 3-4: 60 mg MR orlistat (1 capsule TID), week 5-26: 60 mg MR orlistat (2 capsules TID).
  Arms: MR orlistat
Drug: Conventional orlistat 120 mg, — Orlistat in its conventional form will be Alli® 60 mg during week 1 to 4 and Xenical® 120 mg from week 5 and onwards in matching oral capsules.
  Dosage:
  week 1-2: 60 mg conventional orlistat (1 capsule per day), week 3-4: 60 mg conventional orlistat (1 capsule TID), week 5-26: 120 mg conventional orlistat plus placebo (1 capsule of each TID).
  Other Names: Xenical
  Arms: Conventional orlistat
Drug: EMP16-60/20 — Dosage:
  week 1-2: 60 mg orlistat/20 mg acarbose (1 capsule per day), week 3-4: 60 mg orlistat/20 mg acarbose (1 capsule TID), week 5-26: 60 mg orlistat/20 mg acarbose plus placebo (1 capsule of each TID)
  Arms: EMP16-60/20
Drug: Placebo — Dosage:
  week 1-2: Placebo (1 capsule per day), week 3-4: Placebo (1 capsule TID), week 5-26: Placebo (2 capsules TID)
  Arms: Conventional orlistat; EMP16-60/20; Placebo

SUMMARY:
This is a randomized, double-blind study in participants with overweight or obesity in which the effect of acarbose and the impact of dose on efficacy, safety and tolerability is investigated by comparing the EMP16 combination product with modified release (MR) orlistat, orlistat in its conventional dosage form and placebo.

DETAILED DESCRIPTION:
The study will be conducted at 3 research sites in Sweden. A total of 320 randomized patients are expected to participate in the study for approximately 31 weeks, including a screening period of up to 5 weeks and a 26-weeks treatment period.

EMP16 is indicated for people with obesity with an initial BMI ≥ 30 kg/m² or ≥ 27 kg/m² in the presence of other risk factors (e.g., hypertension, glucose dysregulation and T2DM, and/or dyslipidemia).

Participants will be randomized to either of 5 arms:

* EMP16-120/40, 80 participants
* MR orlistat 120 mg, 80 participants
* Conventional orlistat 120 mg, 80 participants
* EMP16-60/20, 40 participants
* Placebo, 40 participants

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the study.
2. Males or females (sex distribution 50:50, preferably ±5%) aged ≥18 years.
3. BMI ≥ 30 or ≥ 27 kg/m² in the presence of other risk factors based on participant interview e.g., hypertension (either or not treated with antihypertensive agents), glucose dysregulation (defined as elevated fasting glucose ≥6.1 mmol/L or HbA1c >42mmol/mol), Type 2 Ddabetes that is treated with lifestyle changes (no medication allowed), and/or dyslipidemia (either or not treated with antihyperlipidemic agents). If indicated, plasma/serum total cholesterol, LDL, HDL, and/or TGs can be measured to verify eligibility as judged by the Investigator.
4. No clinically significant abnormalities regarding physical examination, vital signs, ECG, and laboratory values at the time of the screening visit, as judged by the Investigator.
5. Adequate renal function: creatinine <1.5 times upper limit of normal (ULN).
6. Adequate hepatic function: aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, gamma-glutamyl transferase <2.5 times upper level of normal (ULN) and bilirubin <1.5 times ULN.

Exclusion Criteria:

1. Weight unstable (≥ 5% reported change during the previous 3 months) preceding screening and randomization.
2. Subjects who are pregnant, who are currently breastfeeding, who intend to become pregnant within the period of the study, or who gave birth within the 6 months preceding the screening visit.
3. Type 2 diabetes treated with medication.
4. History or presence of any clinically significant disease, disorder, or history of surgery which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study including but not limited to:

   * GI problems/diseases, e.g., diseases that affect intestinal absorption and peristalsis such as inflammatory bowel diseases, irritable bowel syndrome (IBS) and Hirschsprung's disease
   * Cholestasis
   * Chronical malabsorption syndrome
   * Severe allergic, cardiac, or hepatic disease
   * Previous GI surgery that might influence GI function significantly, such as previous bariatric surgery, and previous gallbladder surgery as judged by the investigator.

   Potential participants with well-treated chronic diseases (e.g., celiac disease and lactose intolerance) may be included in the study at the discretion of the Investigator.
5. Significant clinical illness within the preceding 2 weeks of the first administration of IMP at the discretion of the Investigator.
6. Any significant medical/surgical procedure or trauma within 4 weeks of the first administration of IMP at the discretion of the Investigator.
7. Any planned major surgery within the duration of the study.
8. Any use of drugs altering glucose metabolism and drugs used for diabetes (A10A and A10B) or drugs that are affected by, or that affect, orlistat and acarbose, within 2 weeks prior to the first administration of IMP.
9. Regular use of prescribed or non-prescribed medication within 2 weeks prior to the first administration of IMP as judged by the Investigator. Patients who are on stable treatment with anti-depressants (e.g., selective serotonin re-uptake inhibitors, SSRI) for at least 2 months can be included at the discretion of the Investigator.
10. Untreated high blood pressure (systolic blood pressure >160 mmHg and diastolic blood pressure >100 mmHg at the screening visit).
11. Known hypersensitivity to any of the test substances.
12. Malignancy within the past 5 years with the exception of in situ removal of basal cell carcinoma.
13. Excessive intake of alcohol, as judged by the Investigator.
14. Current or history of alcohol abuse and/or use of anabolic steroids or drugs of abuse.
15. Positive screen for drugs of abuse, or positive screen for alcohol, at the screening visit (Visit 1).
16. Any positive result at the screening visit (Visit 1) for serum hepatitis B surface antigen, hepatitis C antibody and Human Immunodeficiency Virus (HIV).
17. Plasma donation within 1 month of the screening visit (Visit 1) or any blood donation (or corresponding blood loss) during the 3 months prior to the screening visit.
18. Administration of another new chemical entity (defined as a compound which has not been approved for marketing) or has participated in any other clinical study that included drug treatment within 3 months of the first administration of IMP in this study. Participants consented and screened but not dosed in previous studies are not excluded.
19. Investigator considers the potential participant unlikely to comply with study procedures, restrictions, and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Relative (%) change from baseline in body weight at week 26 | Baseline and week 26
  Efficacy endpoints
Proportion of participants with ≥5% decrease in body weight at week 26 [Please note: This is an FDA required outcome, cannot use "change"] | Baseline and week 26
  Efficacy endpoints

SECONDARY OUTCOMES:
Relative (%) change from baseline in body weight at week 26 (secondary and exploratory comparisons) | Baseline and week 26
  Efficacy endpoints
Proportion of participants with ≥5% (secondary and exploratory comparisons) and ≥10% (all comparisons) decrease in body weight at week 18 and week 26 | Baseline, week 18 and 26
  Efficacy endpoints
Absolute change from baseline in body weight at week 26 | Baseline and week 26
  Efficacy endpoints
Relative (%) change from baseline in body weight during the 26-weeks treatment period | Baseline to week 26
  Efficacy endpoints
Absolute change from baseline in body weight during the 26-weeks treatment period | Baseline to week 26
  Efficacy endpoints
Absolute change from baseline in body mass index (BMI) measured as weight (kg) divided by height (m) squared | Baseline and week 26
  Efficacy endpoints
Absolute change from baseline in waist circumference | Baseline and week 26
  Efficacy endpoints
Absolute change from baseline in sagittal diameter | Baseline and week 26
  Efficacy endpoints
Absolute change from baseline in percentage body fat | Baseline and week 26
  Efficacy endpoints
Absolute change from baseline in Quality of life as measured by the questionnaire Rand-36 (9 different domains) | Baseline and week 26
  Efficacy endpoints
Absolute change from baseline in Quality of life as measured by the questionnaire EQ-5D-5L (measured as one summative value) | Baseline and week 26
  Efficacy endpoints
Absolute change from baseline in self reported meal pattern. Short questionnaire where points are depending on adherence to the Nordic Nutrition recommendations | Baseline and week 26
  Efficacy endpoints.
Absolute change from baseline in self reported sleep, where higher points are given for good sleep duration and good sleep quality | Baseline and week 26
  Efficacy endpoints
Absolute change from baseline in self reported physical activity, where higher points are given for longer duration of moderate and intense physical activity | Baseline and week 26
  Efficacy endpoints
Absolute change from baseline in fasting hemoglobin A1c (HbA1c) | Baseline and week 26
  Efficacy endpoints
Absolute change from baseline in fasting glucose | Baseline and week 26
  Efficacy endpoints
Absolute change from baseline in fasting insulin | Baseline and week 26
  Efficacy endpoints
Absolute change from baseline in fasting total cholesterol | Baseline and week 26
  Efficacy endpoints
Absolute change from baseline in fasting high-density lipoprotein (HDL) | Baseline and week 26
  Efficacy endpoints
Absolute change from baseline in fasting low-density lipoprotein (LDL) | Baseline and week 26
  Efficacy endpoints
Absolute change from baseline in fasting triglycerides (TGs) | Baseline and week 26
  Efficacy endpoints
Absolute change from baseline in fasting Apolipoprotein A1 (ApoA1) | Baseline and week 26
  Efficacy endpoints
Absolute change from baseline in fasting Apolipoprotein B (ApoB) | Baseline and week 26
  Efficacy endpoints
Absolute change from baseline in fasting high sensitivity C-reacting protein (hs-CRP) | Baseline and week 26
  Efficacy endpoints
Absolute change from baseline in fasting albumin | Baseline and week 26
  Efficacy endpoints
Absolute change from baseline in homeostatic model assessment (HOMA) index | Baseline and week 26
  Efficacy endpoints
Absolute change from baseline in Visceral adiposity index (VAI) | Baseline and week 26
  Efficacy endpoints VAI Males = (WC/(39.38+(1.88*BMI)))*(TG/1.03)*(1.31/HDL) VAI Females = (WC/(36.58+(1.89*BMI)))*(TG/0.81)*(1.52/HDL)
Absolute change from baseline in Fatty liver index (FLI) | Baseline and week 26
  Efficacy endpoints. Measured as FLI = 100*e to the power of y /(1+e to the power of y) y= 0.953*ln(TG)+0,139*BMI+0.718*ln(GGT)+0.053*WC-15.3745
Absolute change from baseline in systolic and diastolic blood pressure | Baseline and week 26
  Efficacy endpoints
Absolute change from baseline in heart rate | Baseline and week 26
  Efficacy endpoints
Tolerability, assessed by conventional adverse event (AE) reporting (with special focus on oily spotting and fecal incontinence) | IMP administration until the end-of-study visit. Assessed at all nine visits (both outpatient and telephone visits)
  Safety & tolerability endpoints
Number of withdrawals from study (total and gastrointestinal [GI] related) | Visit 1 until the end-of-study visit. Assessed at all nine visits (both outpatient and telephone visits)
  Safety & tolerability endpoints
Absolute change from baseline in fasting liver enzymes | Baseline and week 26
  Safety & tolerability endpoints (aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase and gamma-glutamyl transferase)

CONTACTS AND LOCATIONS:
Locations (3):
- Sweden (3):
  - CTC Ebbepark, Linköping
  - CTC Karolinska, Solna
  - Clinical Trial Consultants (CTC), Uppsala

IPD SHARING:
Plan to Share IPD: No